CLINICAL TRIAL: NCT05064683
Title: The Effect of Facilitated Tucking and White Noise on Stress and Sleep of Newborns in Nasal CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Yeliz SUNA DAĞ, Researcher assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Yenidoğanlarda uyku
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Newborn; Newborn Sleep; Newborn Stress
Keywords: newborn; sleep; stress; white noise; facilitated tucking
MeSH Terms: interventions — Facilitated Tucking

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- white noise (Experimental): The newborns in the white noise group were listened to white noise for 24 hours using an Mp3 player and a decibel measuring device to measure the sound level.
  Interventions: Other: white noise
- facilitated tucking (Experimental): The newborns in the facilitated tucking were given supine, prone, and lateral positions for 24 hours, depending on their clinical status.
  Interventions: Other: white noise
- control (No Intervention): Newborns in the control group did not receive any treatment other than routine applications while receiving Nasal CPAP support in the neonatal intensive care unit.

INTERVENTIONS:
Other: white noise — Newborns in the control group did not receive any treatment other than routine applications while receiving nasal CPAP support in the neonatal intensive care unit.The newborns in the faciliated tucking group were given supine, prone, and lateral positions for 24 hours, depending on their clinical status.The newborns in the white noise group were listened to white noise for 24 hours using an Mp3 player and a decibel measuring device to measure the sound level.
  Other Names: facilitated tucking; control
  Arms: facilitated tucking; white noise

SUMMARY:
Purpose: Newborns go through biochemical and physiological changes involving all their systems in the first days of their lives and may experience difficulties in adapting to extrauterine life due to various reasons. For newborns whose systems are still immature, leaving the warm, dark, quiet, calm, fluid-filled mother's womb and placing them in the intensive care unit with many stimuli creates intense stress and negatively affects the sleep-wake order necessary for brain development and maturation. Newborns have extensive sleep requirements for the development of their neurosensory system. It is known that the brain activity of newborns in the intrauterine period is similar to the REM (Rapid Eye Movement) sleep activity, and they sleep more than adults and spend most of their sleep in the REM sleep period.Therefore, sleep quality in the newborn period is directly related to healthy development.In this direction, our research was carried out to examine the effects of fetal position and white noise on stress and sleep in newborns with nasal CPAP(Continuous Positive Airway Pressure).

Design and Methods: . This randomized experimental study was conducted on 108 newborns at the gestational week of 26 or higher in the newborn intensive care unit of a university hospital. The researcher applied white noise (n:36), and facilitated tucking(n:36) to the newborns. The control group (n: 36) received no intervention except for the routine clinical practices. Facilitated tucking white noise interventions were applied to the newborns included in study for 24 hours, their stress levels were monitored with the neonatal stress scale, and their sleep durations were monitored with a sleep-wakefulness measurement device and recorded in the newborn follow-up form. Statistical analysis was performed using percentages, means, and ANOVA test.

DETAILED DESCRIPTION:
Sleep is very important for human life and includes both physiological and mental processes in development. Sleep is considered not only as a resting state, but also as a state of intense brain development in which neurotransmitters specific to each sleep stage affect brain maturation. Sleep constitutes a large part of the life of newborns and children. However, total daily sleep time, time to fall asleep, daytime sleep and sleep structure may differ according to the age of the child. It is known that the brain activity of newborns in the intrauterine period is completely similar to the sleep activity of the REM period, and they sleep more than adults and spend most of their sleep in the REM sleep period. Therefore, sleep quality in the newborn period is directly related to healthy development. Newborns who are separated from the warm, dark, quiet, calm, fluid-filled mother's womb, which is the natural environment for them after birth, undergo biochemical and physiological changes involving all their systems in the first days of their life, and may experience difficulties in adapting to extrauterine life due to various reasons. Respiratory problems are among the leading causes of mortality and morbidity in the neonatal period. Nasal CPAP and mechanical ventilation support are the leading techniques used to provide oxygenation and ventilation in the treatment of infants with or without respiratory distress. Nasal CPAP is widely used in newborns, especially preterm infants, both as primary therapy and as a respiratory support method after extubation. However, complications such as hyperemia in the nose, crust formation, bleeding, forehead and face injuries, and infection may develop due to CPAP application. In order to prevent possible complications, neonatal intensive care unit (NICU) nurses should be trained about these risks and complications, specialist nursing care and infection. control protocols should be implemented.Nurses who spend the most time in the neonatal intensive care unit are members of the profession responsible for ensuring the adaptation of newborns to the external environment, optimal growth and development, protection from diseases and maximizing the condition of the newborn, as well as basic nursing practices. The neonatal intensive care nurse monitors the clinical signs and symptoms of the newborn, evaluates and interprets in line with evidence-based information, and determines the care needs with a family-centered approach, makes the nursing diagnosis, plans and implements the care, provides training and counseling . When determining the care needs, it takes into account the risk status of the newborn, the length of hospitalization, the stimuli to which he is exposed, the level of pain and stress, the application of surgical intervention and the presence of invasive applications . In order to prevent situations that reduce or consume the energy resources required for physiological growth of the newborn, to protect the energy resources that are wasted, to accelerate the healing process, to reduce pain, stress, autonomic response and oxygen consumption, to provide sleep pattern, comfort and immobilization, the neonatal intensive care nurse has and non-pharmacological methods. Facilitated tucking white noise are among the non-pharmacological methods frequently used by neonatal nurses.The facilitated tucking is a method that allows the baby to feel and calm down in the womb, to develop behaviors to cope with pain and stress, to feel safe, and to provide body control. In addition, it is a position that improves the sleep pattern that supports motor development, growth and development, and creates a synergistic effect in pain control. It has been reported that this position provides heat and tactile stimulation in newborns, activating the newborns' regulatory systems, preventing painful stimuli from the external environment and reducing the pain experienced by the newborns. Studies have also shown that the facilitated tucking warmth and tactile stimulation in newborns, activates the newborn's own regulatory systems, activates the newborn's attention, prevents painful stimuli originating from the external environment, increases the release of endogenous endorphins, helps the distribution of pain impulses in the spinal cord, and reduces the pain felt by newborn . It has been stated that it is an effective method in reducing the crying time and pain after the procedures.

White noise is a continuous monotonous sound such as the sound of wind, waterfall, ocean waves or rain coming from the environment, and it is a sound that is prepared digitally by mixing different frequency sounds in equal proportions in the laboratory environment and is prepared by calibrating all the frequencies in the sound and it is pleasant to the ear. White noise sources include rain, waterfall, water sounds, hair dryer sound, vacuum cleaner sound, aspirator sound, clock sound, heart sound. When the literature is examined that white noise played during the heel blood collection process in newborns reduces the baby's pain score and shortens the crying time. Similarly, preterm newborns were listened to during the white noise vaccination process and it was found to have a pain-reducing effect compared to the control group.

White noise is similar to the sound in the womb as it is a humming and continuous monotonous sound. It is known that the newborn is affected by the mother's heartbeat while in the womb, and finding this sound and rhythm after birth has a relaxing effect on the newborn. In experimental studies conducted in the relevant field, it has been observed that newborns sleeping in a room where the sound of the uterus is heard fall asleep earlier than those in the room where no sound is heard, and this shows that newborns begin to gain a certain sensitivity to music before they are born.

When the literature is examined, it has been stated facilitated tucking white noise may affect the sleep quality of newborns. However, it has been observed that there is no study examining the difference between facilitated tucking and white noise. In this direction, research was carried out to examine the effects of facilitated tucking and white noise on the stress and sleep of newborns in Nasal CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Patients at 26 and above gestational weeks receiving nasal CPAP support.
* Newborns who do not have a health problem that prevents them from being positioned
* Newborns regularly visited by their mothers in neonatal intensive care clinics

Exclusion Criteria:

* Congenital anomaly of the newborn
* Newborns with hearing loss

Ages: 0 Days to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Changes in sleep | 24 hours
  Nurses followed the sleep duration of newborns with a sleep-wake measurement device for 24 hours and recorded in the Newborn Follow-up Form.

SECONDARY OUTCOMES:
Changes in stress | 24 hours
  Nurses followed their stress levels with the newborn stress scale for 24 hours and recorded them on the newborn follow-up form.Minimum 0 points, 28 maximum 16 points are taken from the scale. As the score increases, the newborns stress level increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

REFERENCES:
- [Background] Çalışır H, Güler F. Yenidoğan Yoğun Bakım Ünitesinde Mekanik Ventilasyon Uygulanan Prematüre Bebeklere Pozisyon Verme.Türkiye Klinikleri J Nurs Sci. 2017;9(3):227-23.2 .
- [Background] Huang YS, Paiva T, Hsu JF, Kuo MC, Guilleminault C. Sleep and breathing in premature infants at 6 months post-natal age. BMC Pediatr. 2014 Dec 16;14:303. doi: 10.1186/s12887-014-0303-6. PMID 25510740
- [Background] Kurt FY, Aytekin A, Çelebi A. 0-3 Yaş Çocuklarda Uyku Sorunlarının Belirlenmesi. Zeynep Kamil Tıp Bülteni. 2018;49(3), 259-263.
- [Background] Küçük S. Yenidoğan yoğun bakım ünitelerinde kaliteli uyku.Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi. 2015; 8(3): 214-217.
- [Background] Arpaci T, Altay N. Yenidoğan Yoğun Bakım Ünitelerinde Bireyselleştirilmiş Gelişimsel Bakım: Güncel Yaklaşımlar. Turkiye Klinikleri Hemşirelik Bilimleri. 2017;9(3): 245-54
- [Background] Başkan AK, Salihoğlu Ö, Tan İ, Akyol B, Hatipoğlu S. İnvaziv Mekanik Ventilatör Desteği Alan Yenidoğanlarda Morbidite ve Mortalite Analizi. Journal of Clinical and Experimental Investigations. 2012; 3 (4): 483-492.
- [Background] Dewez JE, Chellani H, Nangia S, Metsis K, Smith H, Mathai M, van den Broek N. Healthcare workers' views on the use of continuous positive airway pressure (CPAP) in neonates: a qualitative study in Andhra Pradesh, India. BMC Pediatr. 2018 Nov 6;18(1):347. doi: 10.1186/s12887-018-1311-8. PMID 30400844
- [Background] Cakici M, Mutlu B. Effect of Body Position on Cardiorespiratory Stabilization and Comfort in Preterm Infants on Continuous Positive Airway Pressure. J Pediatr Nurs. 2020 Sep-Oct;54:e1-e8. doi: 10.1016/j.pedn.2020.06.015. Epub 2020 Jul 15. PMID 32680615
- [Background] Tiryaki Ö, Çınar N . Devamlı Pozitif Hava Yolu Basıncındaki Yenidoğanın Hemşirelik Bakımı. Turkiye Klinikleri Journal of Nursing Sciences. 2016; 8(1):79-85.
- [Background] Houck CS. Neonatal Pain Management. Pediatric Pain Management for Primary Care, America. 2005, s.361.
- [Background] Ward-Larson C, Horn RA, Gosnell F. The efficacy of facilitated tucking for relieving procedural pain of endotracheal suctioning in very low birthweight infants. MCN Am J Matern Child Nurs. 2004 May-Jun;29(3):151-6; quiz 157-8. doi: 10.1097/00005721-200405000-00004. PMID 15123970
- [Background] Hill S, Engle S, Jorgensen J, Kralik A, Whitman K. Effects of facilitated tucking during routine care of infants born preterm. Pediatr Phys Ther. 2005 Summer;17(2):158-63. doi: 10.1097/01.pep.0000163097.38957.ec. PMID 16357666
- [Background] Axelin A, Salantera S, Lehtonen L. 'Facilitated tucking by parents' in pain management of preterm infants-a randomized crossover trial. Early Hum Dev. 2006 Apr;82(4):241-7. doi: 10.1016/j.earlhumdev.2005.09.012. Epub 2006 Jan 10. PMID 16410042
- [Background] Obeidat H, Kahalaf I, Callister LC, Froelicher ES. Use of facilitated tucking for nonpharmacological pain management in preterm infants: a systematic review. J Perinat Neonatal Nurs. 2009 Oct-Dec;23(4):372-7. doi: 10.1097/JPN.0b013e3181bdcf77. PMID 19915422
- [Background] Huang CM, Tung WS, Kuo LL, Ying-Ju C. Comparison of pain responses of premature infants to the heelstick between containment and swaddling. J Nurs Res. 2004 Mar;12(1):31-40. doi: 10.1097/01.jnr.0000387486.78685.c5. PMID 15136961
- [Background] Johnston CC, Fernandes AM, Campbell-Yeo M. Pain in neonates is different. Pain. 2011 Mar;152(3 Suppl):S65-S73. doi: 10.1016/j.pain.2010.10.008. Epub 2010 Oct 23. PMID 20971562
- [Background] Chorna OD, Slaughter JC, Wang L, Stark AR, Maitre NL. A pacifier-activated music player with mother's voice improves oral feeding in preterm infants. Pediatrics. 2014 Mar;133(3):462-8. doi: 10.1542/peds.2013-2547. Epub 2014 Feb 17. PMID 24534413
- [Background] Kucukoglu S, Aytekin A, Celebioglu A, Celebi A, Caner I, Maden R. Effect of White Noise in Relieving Vaccination Pain in Premature Infants. Pain Manag Nurs. 2016 Dec;17(6):392-400. doi: 10.1016/j.pmn.2016.08.006. Epub 2016 Oct 15. PMID 27751753
- [Background] Standley JM. Music therapy for the neonate. Newborn and Infant Nursing Reviews. 2001;1:211-216.